CLINICAL TRIAL: NCT05457075
Title: Role of Immune Checkpoints in Predicting Response to Neoadjuvant Therapy in Rectal Cancer Patients
Brief Title: Immune Checkpoints in Predicting Response to Neoadjuvant Therapy in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD. PhD, Istanbul Training and Research Hospital
Other Study IDs: Neoadjuvant rectum
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant Therapy; Rectal Cancer; Immune Checkpoints
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma of the rectal cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: Stage II-III rectal cancer patients who have neoadjuvant therapy
  Interventions: Diagnostic Test: Immune checkpoint measure

INTERVENTIONS:
Diagnostic Test: Immune checkpoint measure — The measurement of soluble immune checkpoints of stage II-III rectal cancer before neoadjuvant treatment

SUMMARY:
Colorectal cancer is the third most frequently diagnosed type of cancer in the world. Recent developments in the treatment of cancers suggest that immune checkpoint inhibitors will play an important role. Many studies have documented many types of soluble receptors and ligands that can be detected in plasma in cancer, and plasma levels of these molecules correlate with cancer severity. There is only one study in the literature evaluating the status of soluble immune control points in patients with rectal cancer. The aim of this study is to investigate the role of serum immune checkpoints before neoadjuvant therapy in predicting clinical response in patients with rectal cancer. In this way, it is aimed to show whether immune checkpoints are predictive markers that can predict response to neoadjuvant therapy in patients with stage II-III rectal cancer.

DETAILED DESCRIPTION:
Colorectal cancers are the third most frequently diagnosed cancer type in the world. Recent developments in the treatment of cancers suggest that immune checkpoint inhibitors will play an important role. Among the different immune checkpoint treatments, those containing PD-1 and CTLA-4 stand out as the most effective ones. In clinical trials, anti-CTLA-4 antibody and anti-PD-1 antibody showed great promise by significantly improving overall survival in newly diagnosed and patients who had neoadjuvant treatment against a wide range of solid and hematological malignancies. However, the effects of soluble receptors and ligands on immune system regulation and cancer therapy have been less studied. Soluble receptors and ligands, which are part of a family that includes full-length receptors and ligands, are produced by mRNA expression or cleavage of membrane-bound proteins and are found free in plasma. These structures may play important roles in immune system regulation through interactions between soluble receptors and full-length ligands or between soluble ligands and full-length receptors. Many studies have documented many types of soluble receptors and ligands that can be detected in plasma in cancer patients, and plasma levels of these molecules correlate with cancer severity. As soluble molecules, serum and tissue levels can be easily detected. These molecules are also critical factors for assessing the severity and prognosis of cancer and many other diseases.

In a study, the amounts of PD-L1 and CTLA-4 both on the tumor and soluble in the blood were evaluated, and the high levels of PD-L1 and CTLA-4 were associated with a poor prognosis.

There is only one study in the literature evaluating the status of soluble immune control points in patients with rectal cancer. Of many immune control points, only PD-1 and PD-L1 were evaluated in this study.

In this study, it is planned to include patients who were diagnosed with stage II-III rectal cancer in the General Surgery outpatient clinic of Istanbul Training and Research Hospital between May 2022 and October 2022 and required neoadjuvant treatment in their examinations. Routine rectal cancer surgery will be performed after neoadjuvant treatment of the patients included in the study, and their pathology reports will be examined, and tumor regression scores will be evaluated. Before neoadjuvant treatment, 10 cc of blood will be collected from the patients in a biochemistry tube, their serum will be separated by centrifugation and stored in a -80oC refrigerator. After the collection of all samples, serum immune control points will be evaluated by flow cytometry from the samples.

Thus, it will be determined whether there is any relationship between serum immune checkpoint levels and tumor regression score.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Patients who will receive neoadjuvant therapy with clinically and histopathologically proven stage II-III rectal cancer

Exclusion Criteria:

* Known immunodeficiency
* Having a primary malignancy other than rectal cancer,
* Pregnants,
* Patients younger than 18 years and older than 90 years,
* Patients who refused to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with stage II-III rectal cancer in the General Surgery outpatient clinic of Istanbul Training and Research Hospital between May 2022 and October 2022 and required neoadjuvant treatment
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Soluble immune checkpoints | Before neoadjuvant treatment
  sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Reseach Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tominaga T, Akiyoshi T, Yamamoto N, Taguchi S, Mori S, Nagasaki T, Fukunaga Y, Ueno M. Clinical significance of soluble programmed cell death-1 and soluble programmed cell death-ligand 1 in patients with locally advanced rectal cancer treated with neoadjuvant chemoradiotherapy. PLoS One. 2019 Feb 26;14(2):e0212978. doi: 10.1371/journal.pone.0212978. eCollection 2019. PMID 30807610
- [Result] Sasidharan Nair V, Toor SM, Taha RZ, Shaath H, Elkord E. DNA methylation and repressive histones in the promoters of PD-1, CTLA-4, TIM-3, LAG-3, TIGIT, PD-L1, and galectin-9 genes in human colorectal cancer. Clin Epigenetics. 2018 Aug 6;10(1):104. doi: 10.1186/s13148-018-0539-3. PMID 30081950
- [Result] Omura Y, Toiyama Y, Okugawa Y, Yin C, Shigemori T, Kusunoki K, Kusunoki Y, Ide S, Shimura T, Fujikawa H, Yasuda H, Hiro J, Ohi M, Kusunoki M. Prognostic impacts of tumoral expression and serum levels of PD-L1 and CTLA-4 in colorectal cancer patients. Cancer Immunol Immunother. 2020 Dec;69(12):2533-2546. doi: 10.1007/s00262-020-02645-1. Epub 2020 Jun 23. PMID 32577816